CLINICAL TRIAL: NCT00261820
Title: A Randomized Study To Compare The Safety And Efficacy Of Two Immunosuppressive Regimens In De Novo Renal Allograft Recipients:Sirolimus Plus Mycophenolate Mofetil Plus Corticosteroids Following A Rabbit Anti-Human Thymocyte Globulin Induction (RATG) Vs Tacrolimus Plus Mycophenolate Mofetil Plus Corticosteroids
Brief Title: Study Comparing Two Immunosuppressive Regimens in De Novo Renal Allograft Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468E1-100194
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2006-05-19 (Estimated); Status verified 2006-05

CONDITIONS: Graft Rejection; Kidney Failure; Kidney Transplantation
Keywords: Kidney Transplant
MeSH Terms: conditions — Renal Insufficiency | interventions — Tacrolimus; Mycophenolic Acid; Methylprednisolone; Prednisolone; Sirolimus

INTERVENTIONS:
Drug: tacrolimus
Drug: mycophenolate mofetil
Drug: methylprednisolone
Drug: prednisolone
Drug: sirolimus

SUMMARY:
Evaluate renal graft function (based on the calculated Glomerular Filtration Rate) at 12 months after transplantation in patients receiving either a regimen of sirolimus plus mycophenolate mofetil following an antibody induction (RATG) or a standard regimen combining tacrolimus plus mycophenolate mofetil, both regimens including corticosteroids in patients undergoing renal allograft transplantation. In addition, the two treatment groups will be compared with respect to the incidence of acute rejection at 3, 6 and 12 months following transplantation, and the patient and graft survival at 6 and 12 months after transplantation. The safety of sirolimus plus mycophenolate mofetil following an antibody induction (ATG) will be evaluated beginning in the immediate post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 and < 65 years
* End-stage renal disease, with patients scheduled to receive a primary renal allograft from a cadaveric donor
* Patients receiving a second transplant without an immunological loss of their first graft in the first six months of transplant

Exclusion Criteria:

* Evidence of active systemic or localized major infection at the time of initial sirolimus administration
* Evidence of infiltrate, cavitation, or consolidation on chest x-ray obtained during pre-study screening
* Use of any investigational drug or treatment up to 4 weeks prior to enrollment to the study and during the 12-month treatment phase

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Study Completion 2005-01

PRIMARY OUTCOMES:
- Graft function as measured by Glomerular Filtration Rate (GFR) by Nankivell formula at Month 12 post-
transplantation.

SECONDARY OUTCOMES:
Incidence of occurrence of primary acute rejection biopsy confirmed by a local pathologist using the 1997 Banff
criteria at 3, 6 and 12 Months following transplantation
One year graft biopsy status
Incidence of document infection

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com